CLINICAL TRIAL: NCT03672773
Title: A Phase 2 Study of Continuous Talazoparib Plus Intermittent Low-Dose Temozolomide in Patients With Relapsed or Refractory Extensive-Stage Small Cell Lung Cancer (TRIO-US L-07)
Brief Title: Talazoparib and Low-Dose Temozolomide in Treating Participants With Relapsed or Refractory Extensive-Stage Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Translational Research in Oncology (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001387; NCI-2018-01409 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); TRIO-US L-07 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2018-08-14; First posted 2018-09-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Extensive Stage Small Cell Lung Carcinoma; Refractory Extensive Stage Small Cell Lung Carcinoma
Keywords: Small Cell Lung Cancer; PARP Inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — talazoparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (temozolomide, talazoparib) (Experimental): Participants receive temozolomide PO on days 1-5 and talazoparib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Talazoparib; Drug: Temozolomide

INTERVENTIONS:
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase II trial studies how effective talazoparib and temozolomide are for treating participants with extensive-stage small cell lung cancer that has come back after an initial chemotherapy treatment. Talazoparib, a PARP inhibitor, may stop the growth of tumor cells by preventing them from repairing their DNA. Chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving talazoparib and temozolomide may work better in treating participants with extensive-stage small cell lung cancer than either one alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the efficacy of talazoparib in combination with temozolomide as measured by objective response rate (ORR).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of talazoparib plus temozolomide as measured by progression-free survival (PFS), overall survival, duration of response, and time to response.

II. To evaluate the safety, tolerability of talazoparib plus temozolomide. III. To evaluate the pharmacokinetics of talazoparib when given in combination with temozolomide.

IV. To evaluate patient reported outcomes per the Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).

EXPLORATORY OBJECTIVES:

I. To identify potential biomarkers associated with response to study drug treatment.

OUTLINE:

Participants receive temozolomide orally (PO) on days 1-5 and talazoparib PO once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days and then up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Cytologically or histologically confirmed small cell lung cancer (SCLC) with extensive-stage disease.
* Relapsed (progressed within 6 months) or refractory (progressed during or within 4 weeks of completing 1st line platinum based regimen).
* Measurable disease, as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Archival or fresh tissue biopsy available for exploratory analyses.
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1.
* Able to swallow the study drugs, has no known intolerance to study drugs or excipients, and able to comply with study requirements.
* Female participants of childbearing potential must have a negative pregnancy test at screening and must agree to use a highly effective birth control method (defined in protocol) from the time of the first study drug treatment through 45 days after the last study drug treatment.
* Male participants must use a condom when having sex from the time of the first study drug treatment through 105 days after the last study drug treatment. Contraception should be considered for a non-pregnant female partner of childbearing potential.
* Male and female participants must agree not to donate sperm or eggs, respectively, from the first study drug treatment through 105 days and 45 days after the last study drug treatment, respectively.
* Female participants may not be breastfeeding at baseline through 45 days after the last study drug treatment.
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Glomerular filtration rate (by Cockroft-Gault or equivalent estimation) >= 30 mL/min
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for participants with liver metastases
* Serum total bilirubin =< 1.5 X upper limit or normal (ULN) OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 ULN
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless participant is receiving anticoagulant therapy, as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Has not recovered (recovery is defined as Common Terminology Criteria for Adverse Events (CTCAE) version (v)4 grade =< 1 or return to baseline) from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements.
* Best response of progressive disease per RECIST 1.1 to first-line platinum doublet chemotherapy.
* Has received more than 1 line of cytotoxic therapy

  * Prior immunotherapy and targeted therapies (including rovalpituzumab tesirine) are allowed.
* Prior treatment with a PARP inhibitor (not including iniparib) or temozolomide.
* Use of antineoplastic therapies within 14 days before study treatment initiation.
* Use of any other investigational agent within 14 days before study treatment initiation.
* Received radiation therapy within 14 day before study treatment initiation (single fraction palliative radiotherapy is allowed without a washout).

  * Prior thoracic irradiation and prophylactic cranial irradiation are allowed.
* Major surgery within 14 days before study treatment initiation.
* Diagnosis of myelodysplastic syndrome (MDS).
* Gastrointestinal disorder affecting absorption.
* Current or anticipated use of a prohibited P-gp inhibitor or P-gp inducer or BCRP inhibitors.
* History of another cancer within 2 years before study treatment initiation, with the exception of fully treated cancers unlikely to affect the assessment of the study treatment safety or efficacy including early stage breast, prostate, nonmelanomatous skin, thyroid, cervix and endometrial cancer.
* Any condition (concurrent disease, infection, or comorbidity) that interferes with ability to participate in the study, causes undue risk, or complicates the interpretation of safety data, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate defined as the proportion of participants with a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIS)T 1.1 | Up to 1 year
  Will be provided along with the corresponding exact 2-sided 95% confidence interval calculated using a method based on the F distribution.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) assessed by RECIST 1.1 | From treatment initiation to time of first documentation of objective tumor progression or death on study due to any cause, whichever occurs first, assessed up to 1 year
  Will be summarized for the safety analysis (SA) set. Will be summarized using the Kaplan-Meier method and displayed graphically when appropriate.
PFS assessed by RECIST 1.1 | From treatment initiation to time of first documentation of objective tumor progression or death on study due to any cause, whichever occurs first, assessed up to 1 year
  Will be summarized for the SA set. Will be summarized using the Kaplan-Meier method and displayed graphically when appropriate. Median event times and 2-sided 95% confidence interval for each median will be provided.
Overall survival | From treatment initiation to death by any cause, assessed up to 1 year
  Will be summarized using the Kaplan-Meier method and displayed graphically when appropriate.
Duration of response (CR or PR) per RECIST 1.1 | From the first documentation of objective tumor response, assessed up to 1 year
  Will be summarized using the Kaplan-Meier method and displayed graphically when appropriate.
Time to response (CR or PR) per RECIST 1.1 | From treatment initiation to the first documentation of objective tumor response, assessed up to 1 year
  Will be summarized using the Kaplan-Meier method and displayed graphically when appropriate.
Pharmacokinetics of talazoparib - steady state trough plasma concentrations | Up to 1 year
  To evaluate the pharmacokinetics (steady state trough plasma concentrations) of talazoparib when given in combination with temozolomide

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Goldman, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (6):
- United States (6):
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Orlando Health, Inc. d/b/a Orlando Health UF Health Center, Orlando, Florida
  - Ft. Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Cancer Center of Kansas, Wichita, Kansas